CLINICAL TRIAL: NCT02063087
Title: Shared Decision Making in Parents of Children With Head Trauma: Head CT Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, Davis (Other); University of Minnesota Masonic Children's Hospital (Unknown); Columbia University (Other); Flying Buttress Associates (Unknown); Children's Hospitals and Clinics of Minnesota (Other); Nationwide Children's Hospital (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, M. Fernanda Bellolio, Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-004659; FP00071515 (Other: PCORI)
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Head Injury
Keywords: Head CT; Head Injury; Pediatric; Emergency Department; Decision Aids; Shared Decision Making
MeSH Terms: conditions — Craniocerebral Trauma; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision Aid (Active Comparator): Head CT Decision Aid
  Interventions: Other: Head CT Decision Aid
- Usual Care (No Intervention): Clinicians and patients do not have access to the Head CT Decision Aid

INTERVENTIONS:
Other: Head CT Decision Aid — The decision aid, Head CT Choice, educates parents regarding how the clinician determined the severity of their child's head trauma, their child's quantitative risk for a clinically-important TBI, the pros and cons of cranial CT compared to active observation, and what signs and symptoms parents should watch for in the next 24 hours that should prompt a return visit to the ED.
  Arms: Decision Aid

SUMMARY:
The investigators will test the impact of a decision aid, Head CT Choice, to determine if its use improves parents' knowledge and engagement in decision making and safely decreases healthcare utilization in children presenting to the emergency department with blunt head trauma.

DETAILED DESCRIPTION:
The investigators' long term goal is to promote evidence-based, patient-centered evaluation in the acute setting, to more closely tailor testing to disease risk. The investigators will compare the use of risk stratification tools with usual clinical approaches to treatment selection or administration through the following aim:

Test if the decision aid, Head CT Choice, improves validated patient-centered outcome measures and safely decreases healthcare utilization. The investigators will randomize at the clinician level. Through the use of the intervention, Head CT Choice, the investigators aim to significantly increase parents' knowledge, engagement, and satisfaction, decrease the rate of head CT use, and decrease 7-day total healthcare utilization, with no significant increase in adverse events.

ELIGIBILITY:
Inclusion Criteria:

Parents and their child, seeking care for a child who:

1. Is < 18 years of age;
2. Had blunt trauma above the eyebrows (not isolated to face or eyes);
3. Is positive for at least 1 of the PECARN clinical prediction rule predictors described below:

PECARN Predictors for children < 2 years of age:

Severe mechanism (PECARN definition)* Loss of consciousness > 5 seconds Acting abnormally per parent Initial ED GCS < 15 by attending (or CT decision-maker) Other signs of altered mental status (PECARN definition) Presence of occipital, temporal or parietal scalp hematoma Palpable skull fracture or unclear if skull fracture

PECARN predictors for children 2-18 years of age:

Severe mechanism (PECARN definition)* Any loss of consciousness Any vomiting since the injury Severe headache in ED Initial ED GCS < 15 by attending (or CT decision-maker) Other signs of altered mental status (PECARN definition)** Any sign of basilar skull fracture Clinicians include attending physicians and fellows or midlevel providers caring for children with head trauma

Exclusion Criteria:

Parents of children with:

1. GCS scores < 15
2. Evidence of penetrating trauma, signs of basilar skull fracture, or depressed skull fracture on physical examination
3. Brain tumors
4. Ventricular shunts
5. Bleeding disorder
6. Pre-existing neurological disorders complicating assessment
7. Neuroimaging at an outside hospital before transfer
8. Signs of altered mental status (agitation, somnolence, repetitive questioning, or slow response to verbal communication)
9. Syncope or seizure disorder preceded (led to) head trauma or seizure post head trauma
10. Known to be pregnant
11. Communication barriers such as visual or hearing impairment that may preclude use of the decision aid.
12. Strong suspicion of abuse for this head injury

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 971 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M.Fernanda Bellolio, MD, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - University of California, Davis Medical Center, Sacramento, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of MN, Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospitals and Clincis of MN, St Paul ED, Saint Paul, Minnesota
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Derived] Hess EP, Homme JL, Kharbanda AB, Tzimenatos L, Louie JP, Cohen DM, Nigrovic LE, Westphal JJ, Shah ND, Inselman J, Ferrara MJ, Herrin J, Montori VM, Kuppermann N. Effect of the Head Computed Tomography Choice Decision Aid in Parents of Children With Minor Head Trauma: A Cluster Randomized Trial. JAMA Netw Open. 2018 Sep 7;1(5):e182430. doi: 10.1001/jamanetworkopen.2018.2430. PMID 30646167
- [Derived] Hess EP, Wyatt KD, Kharbanda AB, Louie JP, Dayan PS, Tzimenatos L, Wootton-Gorges SL, Homme JL, Pencille R N L, LeBlanc A, Westphal JJ, Shepel K, Shah ND, Branda M, Herrin J, Montori VM, Kuppermann N. Effectiveness of the head CT choice decision aid in parents of children with minor head trauma: study protocol for a multicenter randomized trial. Trials. 2014 Jun 25;15:253. doi: 10.1186/1745-6215-15-253. PMID 24965659
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Emergency Department Intervention
Arm/Group | Decision Aid | Usual Care
Started | 493 | 478
Completed | 493 | 478
Not Completed | 0 | 0
Period: 7 Day Follow-up
Arm/Group | Decision Aid | Usual Care
Started | 493 | 478
Completed | 493 | 478
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | Usual Care | Total
Number analyzed (Participants) | 493 | 478 | 971
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <2 years old | 123 | 109 | 232
  Age Group: 2 to18 years old | 370 | 369 | 739
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 193 | 396
  Male | 290 | 285 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 62 | 116
  Not Hispanic or Latino | 439 | 416 | 855
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 371 | 347 | 718
  Race: Black | 61 | 54 | 115
  Race: Asian / Pacific Islander / American Indian | 24 | 19 | 43
  Race: Other | 37 | 58 | 95
Region of Enrollment [Number; unit: participants]
  United States | 493 | 478 | 971

OUTCOME MEASURES:

1. Primary Outcome: Assess Parents' Knowledge Regarding Their Child's Risk for a Significant Brain Injury
Description: Knowledge will be measured by means of a post visit survey delivered immediately after the clinical encounter in the emergency department. The investigators will assess parents' knowledge regarding their child's quantitative risk for a significant brain injury, the pros and cons of head CT compared to active observation, and what signs and symptoms parents should watch for in the next 24-48 hours that should prompt a return visit to the ED. Each knowledge question will provide the parent(s) with three options to respond (True, False, or Unsure), and the parent(s) will receive a score of 1 for a correct response and 0 for an incorrect response and any response of 'Unsure' will be considered incorrect. An overall score will be calculated by summing the correct responses and dividing by the number of questions asked.
Time Frame: Day 1 (immediately after the clinical encounter)
Population: Analysis limited to participants with complete data.
Measure: Mean (Standard Deviation); unit: Number of questions correct out of 10
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 467 | 468
Number of questions correct out of 10 | 6.2 (2.0) | 5.26 (2.0)

2. Secondary Outcome: Patient Engagement in the Decision-making Process
Description: Using the OPTION validated scale, the investigators will measure the degree to which clinicians engage parents' in the decision making process. The OPTION scale will be assessed by having 2 observers independently review and score the video recordings of the encounter between the parent and the child's emergency department clinician. The OPTION scale is composed of 12 items with a value of 0-4; they are summed, divided by 48 and multiplied by 100. This creates a score that ranges from 0-100, where higher scores are reflective of a higher level of parental engagement.
Time Frame: Day 1 (during the ED visit)
Population: Analysis limited to patients who consented to recording and had a recording of sufficient quality to analyze
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 266 | 244
Units on a scale | 25 (8.5) | 13.3 (6.5)

3. Secondary Outcome: Decisional Conflict
Description: The investigators will measure the degree of conflict patients experience related to feeling uninformed using the validated Decisional Conflict Scale (DCS). The 16 items of DCS are scored on a 0-4 scale; the items are summed, divided by 16 and then multiplied by 25. The scale is from 0-100 where higher scores are reflective of parental uncertainty about the choice.
Time Frame: Day 1 (immediately after the clinical encounter)
Population: Analysis limited to participants with complete data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 464 | 464
Units on a scale | 14.8 (15.5) | 19.2 (16.6)

4. Secondary Outcome: Trust in the Physician
Description: The investigators will measure parents' trust in their clinician using the validated Trust in Physician Scale (TPS). There are 9 items with a scale of 1-5, the items are subtracted by 1, summed, divided by 9 and then multiplied by 25. The scale ranges from 0-100 where higher values are reflective of higher levels of trust in their physician.
Time Frame: Day 1 (immediately after the clinical encounter)
Population: Analysis limited to patients with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 477 | 469
units on a scale | 91.5 (11.9) | 89.3 (13.7)

5. Secondary Outcome: Parental Satisfaction
Description: The investigators will assess parents' satisfaction by comparing the number of patients who reported being "strongly satisfied" with their choice.
Time Frame: Day 1 (immediately after the clinical encounter)
Population: Analysis limited to participants who completed a post-encounter survey
Measure: Number; unit: participants "Strongly Satisfied"
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 465 | 465
participants "Strongly Satisfied" | 254 | 210

6. Secondary Outcome: Proportion of Children Who Undergo Head CT
Description: The study coordinator will ascertain whether the child underwent head CT in real time and confirm the data by health record review.
Time Frame: Day 1 (anytime during the index emergency department visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 493 | 478
Participants | 109 | 116

7. Secondary Outcome: Healthcare Utilization - Number of Tests Ordered Within 7 Days
Description: The investigators will assess healthcare utilization for the subsequent 7-days after the ED visit. Healthcare utilization will include measures such as hospitalization, re-hospitalization, primary and specialty visits, and diagnostics including CT use which will be obtained via a health record review, review of itemized hospital charges on the UB-92 and UB-04 forms (summary billing statements), and parental report via the 7 day follow-up by the study coordinator. Outcomes are reported as number of tests or procedures per patient, categorized based on the Berenson-Eggers Types of Service (BETOS) codes.
Time Frame: 7-days
Measure: Mean (Standard Deviation); unit: number of tests or procedures performed
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 493 | 478
number of tests or procedures performed
  Evaluation and Management Codes for ED Visit | 1.84 (0.23) | 1.88 (0.2)
  Imaging | 0.65 (0.41) | 0.88 (0.56)
  Tests | 0.41 (0.32) | 0.7 (0.55)
  Procedures | 0.17 (0.13) | 0.26 (0.19)
  Other | 0.23 (0.28) | 0.38 (0.46)
  Unclassified | 0.02 (0.02) | 0.02 (0.03)

8. Secondary Outcome: Rate of Clinically Important Traumatic Brain Injury (ciTBI)
Description: The investigators will assess safety by comparing the rate of ciTBI in each arm of the study. The investigators will define ciTBI as we did in the original PECARN study: death from TBI, intubation for more than 24 hours for TBI, neurosurgical procedure, or hospital admission of 2 nights or more associated with TBI on CT.
Time Frame: 7-days
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 493 | 478
Participants | 0 | 1

9. Secondary Outcome: Fidelity - Options for Care
Description: We will measure the degree to which the intervention is implemented as intended in both intervention and control groups when reviewing the recordings. The recordings in the intervention group will serve as a measure of the fidelity with which the intervention was delivered as intended. We will use a checklist of elements present and absent for quantification of implementation.
Time Frame: Day 1
Population: participants who consented to recording, and with a recording of sufficient quality to be scored
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 267 | 249
Participants
  Decision aid brought into the room | 259 | 0
  Decision aid used during the decision-making | 251 | 0
  Decision aid was used by clinician alone | 89 | 0
  Decision aid was shared with the parent/caregiver | 157 | 0
  Undetermined decision aid use (audio recording) | 5 | 0
  Clinician discuss any options for care | 266 | 233
  Discussed option to get a CT scan now | 257 | 196
  Discussed active observation at home | 260 | 215
  Discussed option to let the ED clinician decide | 14 | 1

ADVERSE EVENTS:
Arm/Group | Decision Aid | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/493 | 0/478
Serious Adverse Events (participants affected / at risk) | 0/493 | 0/478
Other Adverse Events (participants affected / at risk) | 0/493 | 0/478

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No